CLINICAL TRIAL: NCT00513760
Title: Characterization of Transporter Mediated Uptake of Montelukast in Humans
Brief Title: Transporter Mediated Uptake of Montelukast
Acronym: TPORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Edward Mougey, Reserach Scientist, Nemours Children's Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 32711; 32-03215-003 (Other Grant/Funding Number: Nemours internal activity number)
Record Dates: First submitted 2007-08-07; First posted 2007-08-09 (Estimated); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Asthma
Keywords: Pharmacogenetics; Singulair; montelukast; Leukotriene Antagonists; Anti-Asthmatic Agents; Intestinal Absorption; pharmacokinetics; absorption; biochemical transport; Membrane Transport Proteins; Drug Interactions
MeSH Terms: conditions — Asthma | interventions — gatorade

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Coingestion of 240 ml of grapefruit juice with 10 mg of montelukast.
  Interventions: Dietary Supplement: Grapefruit juice
- 2 (Active Comparator): Coingestion of 240 ml of orange juice with 10 mg of montelukast.
  Interventions: Dietary Supplement: Orange Juice
- 3 (Placebo Comparator): Coingestion of 240 ml of Gatorade with 10 mg of montelukast.
  Interventions: Dietary Supplement: Gatorade

INTERVENTIONS:
Dietary Supplement: Grapefruit juice — Coingestion of 240 ml of grapefruit juice with 10 mg of montelukast.
  Other Names: Brand: Great Value frozen concentrated grapefruit juice(Walmart).
  Arms: 1
Dietary Supplement: Orange Juice — Coingestion of 240 ml of orange juice with 10 mg of montelukast.
  Other Names: Brand: Winn Dixie orange juice (Winn Dixie).
  Arms: 2
Dietary Supplement: Gatorade — Coingestion of 240 ml of Gatorade with 10 mg of montelukast.
  Other Names: Brand: Gatorade Rain.
  Arms: 3

SUMMARY:
Leukotriene receptor antagonists (LTRAs) are frequently prescribed to reduce the symptoms associated with asthma. Singulair, manufactured by Merck, is a popular LTRA, however its effectiveness varies greatly between individuals. We are interested in understanding why the effectiveness of Singulair varies so greatly.

For an oral drug such as Singulair to be effective, the body must efficiently absorb it. We have found that blood levels of Singulair vary greatly between individuals, and we think that this variability is responsible for variability in response.

Drug absorption occurs primarily in the intestine. Due to differences in the chemical properties of drugs, some drugs can be absorbed easily while other drugs require help from special proteins produced by the cells that line the intestine. These proteins, or transporters act like turnstiles to allow drugs to move from the intestine to the bloodstream and are known to be inhibited by components of citrus juice. The activity of a transporter can be influenced by individual genetic variability.

We think that Singulair requires help from a transport protein to be absorbed and that genetic variability in this transporter leads to variability in the blood level of Singulair. In this proposal we will use citrus juice (grapefruit and orange) to inhibit intestinal membrane transport proteins and show that Singulair requires these transporters to be efficiently absorbed. Eventually, what we learn from this work will allow doctors to quickly test individuals with asthma to determine how well they will absorb Singulair and possibly other LTRAs. Knowing this will allow the doctor to adjust the drug treatment on an individual basis to maximize benefit in the treatment of asthma.

DETAILED DESCRIPTION:
Montelukast (Merck brand name Singulair) is a selective Cys-LT1 receptor antagonist that is used to control asthma symptoms in children and adults. Although safe and effective, the inter-patient variability in response is substantial (25-60% response rate), which is due in part to genetic variability. For example, we recently reported that polymorphisms in candidate genes that encode proteins in the LT pathway influence responsiveness to the drug.

The long-range goal of our studies is to determine the contribution of genetic variability to the inter-patient variability in montelukast blood levels and responsiveness. In preliminary studies, we found that the plasma concentration vs. time data in single and multiple dose-studies vary more than 10-fold, which could contribute to inter-patient variability in response.

Montelukast is about 64% bioavailable, is cleared by CYP2C9 and CYP3A4 in the liver, and is nearly completely excreted into the bile. The physical properties of montelukast suggest that the drug undergoes transport by solute carrier transporters (SLC family transporters) and/or ATP-binding cassette transporters (ABC family transporters). Recent studies support the idea that genetic variation in genes encoding SLC and ABC transporters can influence the pharmacokinetics of drugs that are substrates for these transporters.

In the present submission, we propose to determine if montelukast is a substrate for SLC and/or ABC transporters. To accomplish this we will coadminister Singulair with citrus juice which contains known inhibitors of membrane transport proteins. If transporters are involved in the absorption of montelukast, then citrus juice should decrease the absorption of montelukast relative to Gatorade. Our working hypothesis for this study is that montelukast is a substrate for SLC (OATP1B3, OATP1B1, OATP2B1, OATP1A2) and ABC (MRP1, MRP2, and MRP3, BCRP) transporters. If true, then the pharmacokinetics of montelukast will be determined by the genetics of the membrane transporters. This highly significant observation will have important implications for understanding the disposition of montelukast in patients, and ultimately will lead to individualization of montelukast therapy in asthma.

ELIGIBILITY:
Inclusion Criteria:

* Doctor diagnosed asthma.
* Must not be taking any medications except for inhaled steroids.

Exclusion Criteria:

* Clinical conditions other than asthma.
* Upper respiratory tract infection within the past 30 days.
* Gastrointestinal conditions.
* Unable to stop taking or are required to begin taking any type of oral medication for the duration of the trial

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2007-06; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Area under the concentration vs. time curve for the serum concentration of montelukast when coingested with grapefruit juice, orange juice, or Gatorade. | Within 12 hours after administration of a single 10 mg dose.

SECONDARY OUTCOMES:
Improvement in respiratory function as assessed by spirometry, and impulse oscillometry vs. serum concentration of montelukast. | Within 12 hours after administration of a single 10 mg dose.

CONTACTS AND LOCATIONS:
Overall Officials: Edward B Mougey, Ph.D., Principal Investigator — Nemours Children's Clinic
Locations (1):
- Nemours Children's Clinic, Jacksonville, Florida, United States

REFERENCES:
- [Background] Lima JJ. Treatment heterogeneity in asthma: genetics of response to leukotriene modifiers. Mol Diagn Ther. 2007;11(2):97-104. doi: 10.1007/BF03256228. PMID 17397245
- [Background] Lima JJ, Zhang S, Grant A, Shao L, Tantisira KG, Allayee H, Wang J, Sylvester J, Holbrook J, Wise R, Weiss ST, Barnes K. Influence of leukotriene pathway polymorphisms on response to montelukast in asthma. Am J Respir Crit Care Med. 2006 Feb 15;173(4):379-85. doi: 10.1164/rccm.200509-1412OC. Epub 2005 Nov 17. PMID 16293801
- See also: Merck's Singulair site — http://www.singulair.com/